CLINICAL TRIAL: NCT07220876
Title: A Prospective, Multicenter, Single-Arm, Open-Label Clinical Trial of the Safety and Effectiveness of the VisiPlate Aqueous Shunt in Patients With Refractory Open-Angle Glaucoma
Brief Title: Safety and Effectiveness of the VisiPlate Aqueous Shunt in Patients With Refractory Open-Angle Glaucoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Avisi Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP0005
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Open Angle Glaucoma (OAG)
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Device: VisiPlate Glaucoma Implant

INTERVENTIONS:
Device: VisiPlate Glaucoma Implant — Implant (micro-shunt) for glaucoma patients

SUMMARY:
A Prospective, Multicenter, Single-Arm, Open-Label Clinical Trial

DETAILED DESCRIPTION:
To evaluate the safety and effectiveness of VisiPlate Aqueous Shunt to lower intraocular pressure (IOP) in subjects with open-angle glaucoma for whom medical and surgical treatments have failed.

ELIGIBILITY:
Inclusion Criteria:

* Open angle, pseudoexfoliative or pigmentary glaucoma
* IOP at preoperative visit of ≥ 20mmHg and ≤ 40mmHg
* Visual field mean deviation score of -3dB or worse
* Area of healthy, free and mobile conjunctiva in the target quadrant
* Shaffer angle grade ≥ 2 in the target quadrant

Exclusion Criteria:

* Angle closure glaucoma
* Congenital, neovascular or other secondary glaucomas
* Previous intraocular surgery, with the exception of uncomplicated cataract surgery
* Previous glaucoma shunt/valve in the target quadrant
* Clinically significant inflammation or infection in the study eye within 30 days prior to the operative visit
* History of corneal surgery, corneal opacities or corneal disease
* Retinal or optic nerve disorders, either degenerative or evolutive, that are not associated with the existing glaucoma condition

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects (eyes) achieving a ≥ 20% reduction in mean diurnal intraocular pressure | 12 Months
  The eye is filled with a special fluid. The intraocular pressure is the amount of fluid that builds up in the eye. The primary outcome is the number of people whose eye pressure went down by at least 20%.

SECONDARY OUTCOMES:
Percentage change in mean diurnal IOP | 12 months
  How much the average eye pressure during the day went up or down, shown as a percent.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (10):
  - Arizona Advanced Eye Research, Glendale, Arizona
  - Sacramento Eye Consultants, Sacramento, California
  - ICON Eye Care, Grand Junction, Colorado
  - Mile High Eye Institute, Sheridan, Colorado
  - Cleveland Clinic- Cole Eye Institute, Cleveland, Ohio
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Glaucoma Associates of Texas, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - The Eye Centers of Racine & Kenosha, Kenosha, Wisconsin
- South Africa (2):
  - Lynette Venter, Bloemfontein
  - Pretoria Eye Institute, Pretoria

IPD SHARING:
Plan to Share IPD: No